CLINICAL TRIAL: NCT03872635
Title: Effects of Drug or Drink Intervention and Temperature Protectionon for Cervical Cancer Patients on Insulin Resistance and Tumor Immunity
Brief Title: Effects of Anesthesia on Tumor Immunity and Insulin Resistance During Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJCAAN01
Record Dates: First submitted 2019-02-23; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Cervical Cancer; Carbohydrate; Tumor Immunity
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHO Drinking Grope (Experimental): receive 300mL of an oral carbohydrate liquid supplement 2 hour before surgery
  Interventions: Other: oral carbohydrate liquid
- Traditional fast Grope (No Intervention): fast on standard hospital protocol (8 hour fasting for solid and 4 hour fasting for clear liquid

INTERVENTIONS:
Other: oral carbohydrate liquid — patients undergoing neoadjuvant chemotherapy and radical hysterectomy with bilateral pelvic lymph node dissection were randomized to receive 300mL of an oral carbohydrate liquid supplement 2 hour before surgery
  Arms: CHO Drinking Grope

SUMMARY:
To evaluate the effects of preoperative oral carbohydrate on postoperative insulin resistance and tumor immunity in cervical cancer patients with neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Fifty-one patients undergoing neoadjuvant chemotherapy and radical hysterectomy with bilateral pelvic lymph node dissection were randomized to receive 300mL of an oral carbohydrate liquid supplement 2 hour before surgery(CHO group) or to fast on standard hospital protocol (8 hour fasting for solid and 4 hour fasting for clear liquid)(FAST group).According to inclusion and exclusion standards, twenty-six patients undergoing the same surgery and standard fasting were selected as control group. Baseline and postoperative measurements of insulin sensitivity were assessed in term of fasting plasma glucose(FPG),fastingainsulin(FINS),HOMA-insulinaresistance(HOMA-IR),HOMA-insulin secretion function index(HOMA-IX) , HOMA-beta cell function index(HOMA-β),serum C-peptide and glucagon.Baseline and postoperative measurements of tumor immunity were evaluated using NK cell and T-cell dynamics.VAS score was introduced to assess preoperative comfort.

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged from 18 to 60 years old were ASA level I to II, and the informed consent was signed by the patients, which was approved by the ethics committee of the hospital.
2. Cervical squamous cell carcinoma was confirmed by cervical biopsy before pathologic surgery. CT showed no distant metastasis. All patients underwent total hysterectomy, bilateral adnexectomy and pelvic lymph node dissection.
3. Fasting blood glucose was normal without diabetes, impaired glucose tolerance or other metabolic diseases.
4. no gastric emptying dysfunction.

Exclusion Criteria:

1. Dabetes
2. Patients with obstruction of gastric emptying, such as pyloric obstruction, gastroesophageal reflux, nausea and vomiting, etc
3. Obese (BMI >32) or severely malnourished (BMI<18.5)
4. Distant metastasis, multiple primary cancers and recurrent tumors
5. Patients with functional disorders of respiratory system, circulatory system, immune system, nervous system, urinary system and other organs
6. Received blood transfusion and nutritional support within 2 weeks before surgery
7. The supplement contains the sugar solution, the blood transfusion, the application glucocorticoid, the sympathetic blood vessel activity medicine in the operation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
insulin resistance | in 24 hrs
  The patient's insulin resistance was determined by fasting plasma glucose(FPG),fastingainsulin(FINS), andHOMA-IR=FPG（mmol/L）×FINS（mIU/L）/22.5

SECONDARY OUTCOMES:
tumor immunity | in 24 hrs
  The patient's tumor immune level was determined by changes in T cells (CD3+、CD4+、CD8+、CD44+) and NK cells in the patient's blood

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fuqing Zhang, Fuzhou, Fujian
  - Mengxia Yao, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang F, Yao M, Lin Z, Chen Y, Jiang H, Zeng M, Chen W. The Effects of Preoperative Oral Carbohydrate on Frequency of T and NK Cells in Patients with Cervical Cancer Treated Using Neoadjuvant Chemotherapy and Surgery: A Prospective Cohort Study. Biomed Res Int. 2020 Mar 16;2020:2101480. doi: 10.1155/2020/2101480. eCollection 2020. PMID 32309426